CLINICAL TRIAL: NCT04118452
Title: A Randomized, Controlled Trial of a Telephone-Based Developmental Care Coordination System
Brief Title: Achieving My Potential: A Randomized, Controlled Trial of a Telephone-Based Developmental Care Coordination System
Acronym: AMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Kaiser Permanente School of Medicine (Other); Virginia Commonwealth University (Other); Information and Referral Federation of Los Angeles County (211 LA County) (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Paul Chung, Adjunct Professor of Pediatrics and Health Policy & Management, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-001556; 7R01HD092406-02 (NIH)
Record Dates: First submitted 2019-09-30; First posted 2019-10-08 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Child Development; Health Services Research
Keywords: early childhood development; developmental screening; care coordination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention + Usual Care + Developmental Screening Results (Experimental): Intervention group families will receive usual care and developmental screening results will be shared with each child's primary care provider. In addition, they will be connected via telephone to 2-1-1 prior to their scheduled well-child visit for the telephone-based early childhood development care coordination intervention.
  Interventions: Behavioral: Telephone-based early childhood developmental care coordination
- Usual Care + Developmental Screening Results (No Intervention): This group will receive usual care. In addition, developmental screening results will be shared with each child's primary care provider.

INTERVENTIONS:
Behavioral: Telephone-based early childhood developmental care coordination — The 211LA care coordinator will review developmental screening results and provide referral recommendations to the family and use 211LA's extensive resource directory and agency relationships to identify appropriate referrals. The 211LA care coordinator will provide a report to the clinical provider containing recommendations for follow-up and a care coordination plan. The report will be scanned into the EMR (Electronic Medical Record) by clinic staff and be available for provider review. The 211LA care coordinator will also make all recommended referrals and will call the family monthly until 1) children begin receiving services, 2) families refuse services, or 3) children are deemed ineligible by service providers.
  Arms: Intervention + Usual Care + Developmental Screening Results

SUMMARY:
The proposed project is a randomized controlled trial of a telephone-based early childhood developmental care coordination system, in partnership with 2-1-1 Los Angeles County (211LA), part of a national network of 2-1-1 call centers covering 93% of the US population. The study will test the effectiveness of 211LA in increasing referrals for developmental evaluation, increasing the numbers of children deemed eligible for services, and increasing the number of children actually receiving interventions.

DETAILED DESCRIPTION:
The trial will enroll 662 children ages 1-3 years who receive well-child care at one of 10 partner clinic sites (belonging to 4 partner clinic systems). The research study team will conduct developmental screening on all children using the Parental Evaluation of Developmental Status (PEDS) Online system, and randomize children 1:1 into intervention (connection to 211LA for developmental care coordination + usual care) or control (usual care alone, with developmental care coordination conducted by clinic staff).

Primary outcomes will include referrals to early intervention evaluations, eligibility for intervention services, and receipt of services. The investigators will measure these outcomes through parent report, medical record review, and 211LA data, at 6 months after enrollment. For children with elevated developmental risk based on the PEDS Online results, the study will assess development using the PEDS:DM-AL (Parents' Evaluation of Developmental Status: Developmental Milestones - Assessment Level), conducted at baseline as well as 12 and 24 months after enrollment. For all children, research study team personnel will administer the language subscale of the PEDS:DM-AL at baseline, 12 months and 24 months, to evaluate development over time in the two groups. The investigators will measure behavioral outcomes for all children using the externalizing behavior subscale of the Child Behavior Checklist.

Expected findings include higher rates of referrals, eligibility, and receipt of intervention services among intervention group participants, and greater developmental gains among children in the intervention group. The study will also examine the costs of the program in relation to these outcomes, to estimate the costs and potential long-term benefits of this model. If effective, the model has the potential to disseminate rapidly throughout the 2-1-1 network and transform developmental care coordination in the US.

ELIGIBILITY:
Inclusion Criteria:

* A patient in one of the four partner community clinic systems (ChapCare, Kaiser Permanente LA Medical Center, South Central Family Health Center, and Via Care)
* A patient with an upcoming one- to three-year old well child appointment scheduled
* Child aged 11-42 months

Exclusion Criteria:

* Parent who does not speak English or Spanish
* Child with history of developmental and/or behavioral diagnosis or having been referred to or received developmental and/or behavioral services.
* Child has a sibling already enrolled in the study.

Ages: 11 Months to 42 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 565 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Chung, MD MS, Principal Investigator — Kaiser Permanente School of Medicine
Locations (4):
- United States (4):
  - South Central Family Health Center, Los Angeles, California
  - Via Care, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - ChapCare, Pasadena, California

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared within 2 years of study completion.
Access Criteria: Proposals should be directed to paul.j.chung@kp.org. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website, to be provided when requests are approved.

REFERENCES:
- [Background] Nelson BB, Thompson LR, Herrera P, Biely C, Arriola Zarate D, Aceves I, Estrada I, Chan V, Orantes C, Chung PJ. Telephone-Based Developmental Screening and Care Coordination Through 2-1-1: A Randomized Trial. Pediatrics. 2019 Apr;143(4):e20181064. doi: 10.1542/peds.2018-1064. PMID 30894408

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention + Usual Care + Developmental Screening Results: Intervention group families will receive usual care and developmental screening results will be shared with each child's primary care provider. In addition, they will be connected via telephone to 2-1-1 prior to their scheduled well-child visit for the telephone-based early childhood development care coordination intervention.
  Telephone-based early childhood developmental care coordination: The 211LA care coordinator will review developmental screening results and provide referral recommendations to the family and use 211LA's extensive resource directory and agency relationships to identify appropriate referrals. The 211LA care coordinator will provide a report to the clinical provider containing recommendations for follow-up and a care coordination plan. The report will be scanned into the EMR by clinic staff and be available for provider review. The 211LA care coordinator will also make all recommended referrals and will call the family monthly until 1) children begin receiving services, 2) families refuse services, or 3) children are deemed ineligible by service providers.
Period: Overall Study
Arm/Group | Intervention + Usual Care + Developmental Screening Results | Usual Care + Developmental Screening Results
Started | 282 | 283
6 Month Survey | 249 | 263
12 Month Survey | 251 | 256
24 Month Survey | 250 | 249
Completed (Completed 12 Month or 24 Month Follow-Up Survey) | 260 | 261
Not Completed | 22 | 22
Not completed — Lost to Follow-up | 5 | 5
Not completed — Withdrawal by Subject | 17 | 17

BASELINE CHARACTERISTICS:
Population: 565 participants were enrolled in the study and 559 completed the baseline survey, including demographic information.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention + Usual Care + Developmental Screening Results | Usual Care + Developmental Screening Results | Total
Number analyzed (Participants) | 278 | 281 | 559
Age, Continuous [Mean (Standard Deviation); unit: Months] | 19.4 (8.1) | 20.6 (8.7) | 20.0 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 123 | 247
  Male | 154 | 158 | 312
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 241 | 235 | 476
  Not Hispanic or Latino | 37 | 45 | 82
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 7 | 8 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 5 | 13
  White | 63 | 60 | 123
  More than one race | 30 | 41 | 71
  Unknown or Not Reported | 168 | 163 | 331
Region of Enrollment [Number; unit: participants]
  United States | 278 | 281 | 559

OUTCOME MEASURES:

1. Primary Outcome: Referral to, Eligibility for, and Receipt of Early Childhood Developmental Services 6 Months After Enrollment
Description: The primary outcome will be assessed by 1) the percentage of children who are successfully referred to early childhood service organizations for evaluation, and 2) the percentage of children who receive services.
Time Frame: 6 months after enrollment
Measure: Number; unit: percentage of children
Arm/Group | Intervention + Usual Care + Developmental Screening Results | Usual Care + Developmental Screening Results
Number analyzed (Participants) | 249 | 263
percentage of children
  Received a referral to early childhood developmental services | 24.5 | 16.3
  Received early childhood developmental services | 14.5 | 8.8

2. Primary Outcome: Child Developmental Outcomes
Description: The PEDS:DM-AL (Parents' Evaluation of Developmental Status: Developmental Milestones - Assessment Level) is an assessment measure of development, social-emotional, and behavioral health that provides age-equivalent and percent delay scores for each domain measured. The domains included in the full assessment are: fine motor, gross motor, expressive language, receptive language, self-help, social-emotional, and academic/pre-academic, and cognitive. This study utilizes the expressive language and receptive language domains to measure child developmental outcomes. This measure will be reported as a Rough Standard Score (RSS), the child's "developmental age" as shown by the tool divided by their actual age. A score of 100 means the child is scored by the instrument as being where we would expect developmentally given their age; lower scores mean the child is developmentally delayed, and higher scores mean the child is ahead of the curve.
Time Frame: Baseline and 24 months after enrollment
Measure: Mean (Standard Deviation); unit: Standardized Score
Arm/Group | Intervention + Usual Care + Developmental Screening Results | Usual Care + Developmental Screening Results
Number analyzed (Participants) | 250 | 249
Standardized Score
  PEDS DM-AL Expressive Language Standardized Score - Baseline | 125.3 (41.3) | 125.4 (40.6)
  PEDS DM-AL Expressive Language Standardized Score - 24 Months | 119.2 (35.6) | 117.6 (41.2)
  PEDS DM-AL - Receptive Language Standardized Score - Baseline | 123.6 (55.9) | 124.0 (50.4)
  PEDS DM-AL Receptive Language Standardized Score - 24 Months | 139.2 (48.8) | 137.3 (50.1)

3. Secondary Outcome: Number of Children Who Have Received Referrals and Number of Children Who Have Received Services
Description: The secondary outcome will be assessed by the number of 1) children with referrals made, and 2) children with services received; the investigators will primarily consider referrals to high-level intervention services for developmental and behavioral problems, but will also track referrals to development-related preventive and support services.
  Intervention services include Part C early intervention (EI), Part B early childhood special education (ECSE), physical therapy (PT), occupational therapy (OT), and speech therapy.
  Early care and education (ECE) includes child care, preschool, Head Start, and Early Head Start.
Time Frame: 6 months after enrollment
Measure: Number; unit: participants
Groups:
- High or Moderate Risk - Intervention + Usual Care + Developmental Screening Results: Intervention group families will receive usual care and developmental screening results will be shared with each child's primary care provider. In addition, they will be connected via telephone to 2-1-1 prior to their scheduled well-child visit for the telephone-based early childhood development care coordination intervention.
  Telephone-based early childhood developmental care coordination: The 211LA care coordinator will review developmental screening results and provide referral recommendations to the family and use 211LA's extensive resource directory and agency relationships to identify appropriate referrals. The 211LA care coordinator will provide a report to the clinical provider containing recommendations for follow-up and a care coordination plan. The report will be scanned into the EMR by clinic staff and be available for provider review. The 211LA care coordinator will also make all recommended referrals and will call the family monthly until 1) children begin receiving services, 2) families refuse services, or 3) children are deemed ineligible by service providers.
  This is a subgroup of children enrolled in the intervention who, at baseline, were determined to have a moderate or high risk for developmental delay.
- High or Moderate Risk - Usual Care + Developmental Screening Results: This group will receive usual care. In addition, developmental screening results will be shared with each child's primary care provider.
  This is a subgroup of children enrolled in usual care who, at baseline, were determined to have a moderate or high risk for developmental delay.
Arm/Group | Intervention + Usual Care + Developmental Screening Results | High or Moderate Risk - Intervention + Usual Care + Developmental Screening Results | Usual Care + Developmental Screening Results | High or Moderate Risk - Usual Care + Developmental Screening Results
Number analyzed (Participants) | 249 | 83 | 263 | 95
participants
  Received a referral for intervention services | 61 | 47 | 43 | 32
  Received intervention services | 36 | 30 | 23 | 16
  Received a referral for early care and education (ECE) services | 144 | 49 | 40 | 16
  Received early care and education (ECE) services | 65 | 30 | 27 | 9

ADVERSE EVENTS:
Time Frame: 2 years
Description: This research study is considered minimal risk and was conducted with participants who were healthy children recruited from usual care at health clinics. As such, they were not at risk for all-cause mortality, serious adverse events, or other adverse events.
Arm/Group | Intervention + Usual Care + Developmental Screening Results | Usual Care + Developmental Screening Results
All-Cause Mortality (participants affected / at risk) | 0/278 | 0/281
Serious Adverse Events (participants affected / at risk) | 0/278 | 0/281
Other Adverse Events (participants affected / at risk) | 0/278 | 0/281

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/52/NCT04118452/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT04118452/ICF_001.pdf